CLINICAL TRIAL: NCT04742231
Title: Use of Handheld Dynamometer As a Novel Tool to Assess Motor Function During Awake Craniotomy for Brain Lesions Located Within or Adjacent to the Motor Cortex: a Single-Center Pilot Study
Brief Title: Handheld Dynamometer During Awake Craniotomy Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kaisorn L. Chaichana, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: 20-004730
Record Dates: First submitted 2020-12-16; First posted 2021-02-08 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Brain Lesion; Brain Tumor Adult; Brain Tumor
Keywords: Awake Craniotomy; Dynamometer; Motor; Brain Mapping
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Cohort 1. Patients with brain lesions in non-motor areas undergoing an awake craniotomy (AC) (Experimental): 5 patient minimum
  Interventions: Device: Hand-held dynamometer
- Cohort 2. Patients with brain lesions within or proximal to motor areas undergoing an AC (Experimental): 5 patient minimum
  Interventions: Device: Hand-held dynamometer

INTERVENTIONS:
Device: Hand-held dynamometer — Maximum Grip Strength will be measured using a hand-held dynamometer (K-FORCE Grip dynamometer®. Kinvent Biomequanique S.A.S, Montpellier, France) during the preoperative, intraoperative (Awake craniotomy) and postoperative period.

SUMMARY:
The primary purpose of this study is to assess the feasibility, safety and reliability of the use of handheld dynamometry in evaluating intraoperative motor function for patients undergoing awake craniotomy for the resection of brain lesions located within or adjacent to the motor cortex.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old.
* Primary or Recurrent Brain tumors
* Single brain lesion
* Lesion within or adjacent to the motor cortex- Lesion located within the primary or supplementary motor area (Verified by preoperative fMRI and DTI).

Exclusion Criteria:

* Patients < 18 years old.
* Major comorbidities (congestive heart failure, severe chronic obstructive pulmonary disease, morbid obesity, obstructive sleep apnea).
* Patients with cognitive, intellectual or psychiatric impairment that could affect the capacity of following instructions evaluated during preoperative neuropsychological testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
Intraoperative maximum grip strength (KgF) baseline | 1 day
  Maximum grip strength (KgF) will be measured using hand-held dynamometry every 2 minutes from the time the patient awakes until the end of surgery. Intraoperative maximum grip strength baseline is defined as the mean of 3 consecutive measures with <10% variability.
Intraoperative maximum grip strength (KgF) variability | 1 day
  To validate the use of hand-held dynamometry as an adequate tool to monitor intraoperative motor function during awake craniotomies (AC), maximum grip strength (KgF) will be measured every 2 minutes from the time the patient awakes to the end of surgery. The intra-individual variability will be defined as the percent difference between sets with 10% or greater defined as substantial variability.
Maximum grip strength (KgF) variability from preoperative baseline | 1 day
  To validate the use of hand-held dynamometry as an adequate tool to monitor intraoperative motor function during AC, each patient will be baselined (mean of 6 consecutive measurements) during the preoperative neuropsychology evaluation. Variability from preoperative baseline will be calculated as a percentile [ (Preoperative Baseline/ Intraoperative Baseline)/ Preoperative Baseline) * 100]
Operative Time (Minutes) | 1 day
  Defined as the duration of the procedure from the initiation of skin incision to the completion of skin closure according to anesthesia records. Measured in minutes.

SECONDARY OUTCOMES:
Correlation Coefficient (ρ) between hand-held dynamometry and manual motor testing during AC | 1 day
  Concordance between hand-held dynamometer and manual motor testing will be evaluated using Spearmans' correlation coefficient.
Postoperative Maximum Grip Strength (KgF) | 1 month
  Postoperative Maximum Grip strength (KgF) will be measured using hand-held dynamometer at day 1 and at 1 month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Kaisorn Chaichana, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials